CLINICAL TRIAL: NCT01518023
Title: Long Term Diabetes Improvement After Cancer Gastrectomy and Colectomy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Joel Faintuch, Associate Professor, Department of Gastroenterology, University of Sao Paulo
Other Study IDs: Lessdiabetes
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes Mellitus; Prediabetes; Morbid Obesity; Gastric Cancer; Colorectal Cancer
Keywords: diabetes mellitus; prediabetes; fasting blood glucose; HbA1c; Roux en Y gastric bypass; Cancer gastrectomy; Cancer colorectal surgery
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Obesity, Morbid; Stomach Neoplasms; Colorectal Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cancer gastrectomy: Patients previously submitted to partial/total gastrectomy for gastric cancer
  Interventions: Other: Interview, questionnaire, updated biochemical tests
- Colorectal cancer operation: Patients previously submitted to right colectomy or rectosignoidectomy for cancer
  Interventions: Other: Interview, questionnaire, updated biochemical tests
- Bariatric patients: Morbidly obese participants who underwent antiobesity Roux-en-Y gastric bypass
  Interventions: Other: Interview, questionnaire, updated biochemical tests

INTERVENTIONS:
Other: Interview, questionnaire, updated biochemical tests — Patients will be interviewed and questioned about nutritional status, diet, drugs and diagnosis/clinical course of diabetes. Routine biochemical tests will be searched and if necessary updated.

SUMMARY:
There is evidence that gastrointestinal operations for non weight-losing purposes are beneficial for diabetes mellitus. Aiming to analyze such hypothesis, patients submitted to gastric bypass for morbid obesity, gastrectomy for gastric cancer and colectomy for colo-rectal cancer will be compared. The end point will be changes in fasting blood glucose and hemoglobin A1c concentration.

DETAILED DESCRIPTION:
In a prospective protocol with retrospective information, patients (N=240) undergoing bariatric Roux-en-Y gastric bypass (n=80), cancer subtotal or total gastrectomy (n=80) and right colectomy or rectosigmoidectomy (n=80) with follow-up >3 years free of disease, with or without previously impaired fasting blood glucose, will be recruited. Patients will be submitted to a questionnaire involving diet, diagnosis of diabetes and glucose-lowering drugs, body weight and other clinical items. Preoperative information available in the hospital system will be completed and current findings will be updated, including body mass index and biochemical measurements. Using the outcomes of the bariatric population as benchmark, both concerning diabetics that were ameliorated and nondiabetics that progressed to new-onset diabetes,results in the other groups will be compared. The study should answer whether gastric and colorectal surgery for cancer 1) Are beneficial for established diabetes; 2) Attenuate the conversion of normal patients to diabetes, both within a follow-up period of 3- 12 years;

ELIGIBILITY:
Inclusion Criteria:

* Follow-up period > 3 years,
* weight stable in the last year

Exclusion Criteria:

* Reoperation or take-down of original operation,
* consumptive diseases,
* protein-calorie malnutrition,
* organ failures,
* pancreatic surgery,
* cell or organ transplantation,
* type 1 diabetes,
* cognitive impairment or Alzheimer disease,
* refusal to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females submitted to elective curative operations will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose | 3-12 years change
  Glucose improvement or deterioration comparing preoperative versus late postoperative value. Classification according to the American Diabetes Association

SECONDARY OUTCOMES:
HbA1c | 3-12 years
  Same as fasting blood glucose (preoperative versus current change). Classification according to the American Diabetes Association.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Faintuch, MD, PhD, Study Chair — Hospital das Clinicas, Sao Paulo, Brazil
Locations (1):
- Hospital das Clinicas- Central Institute ICHC- 9th Floor Rm 9077, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Faintuch J, Yamaguchi CM, Dias MC, Santo MA, Faintuch JJ, Cecconello I. Biochemical correlates of bariatric-responsive diabetes. Diabetes Technol Ther. 2010 Sep;12(9):707-15. doi: 10.1089/dia.2010.0018. PMID 20707737
- [Background] Kim JW, Cheong JH, Hyung WJ, Choi SH, Noh SH. Outcome after gastrectomy in gastric cancer patients with type 2 diabetes. World J Gastroenterol. 2012 Jan 7;18(1):49-54. doi: 10.3748/wjg.v18.i1.49. PMID 22228970
- [Derived] Hayashi SY, Faintuch J, Yagi OK, Yamaguchi CM, Faintuch JJ, Cecconello I. Does Roux-en-Y gastrectomy for gastric cancer influence glucose homeostasis in lean patients? Surg Endosc. 2013 Aug;27(8):2829-35. doi: 10.1007/s00464-013-2829-3. Epub 2013 Feb 23. PMID 23436087